CLINICAL TRIAL: NCT01460784
Title: Changes in Adipokines and Adiposity During Puberty and Young Adulthood
Brief Title: STAGES Trial: Study of Adiposity, Growth and Endocrine Stages
Acronym: STAGES
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nicole L. Mihalopoulos, Associate Professor of Pediatrics, University of Utah
Other Study IDs: IRB_00031720; 1K23HL092069-01A2 (NIH)
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
Keywords: Metabolic dysfunction; Insulin resistance; Brown adipose tissue; Dyslipidemia
MeSH Terms: conditions — Obesity; Insulin Resistance; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buffy coat in -80F long-term storage
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- N=60: Cross-sectional study of obese young adults who underwent PET/CT after cold exposure to identify active brown fat. No intervention. Enrolled 44 participants.
- N=600: Cross-sectional study of patients undergoing clinical PET/CT to identify active brown fat. No intervention. Enrolled 405 participants.
- N=220: Longitudinal observational study of obese adolescents to determine changes in adiposity and adipokines during puberty. No intervention. Enrolled 125 participants.

SUMMARY:
The investigators propose to conduct a cross-sectional study of 60 participants who are 18-30 years of age to undergo research PET/CT. The purpose of this study is to investigate the relationships between Brown Adipose Tissue (BAT), the adiponectin/leptin (A/L) ratio, and components of the metabolic syndrome in young adults.

DETAILED DESCRIPTION:
We propose to conduct a cross-sectional study of 60 participants who are 18-30 years of age to undergo research PET/CT. The purpose of this study is to investigate the relationships between Brown Adipose Tissue (BAT), the adiponectin/leptin (A/L) ratio, and components of the metabolic syndrome in young adults. This study is part of a larger study aimed at understanding the mechanism of brown adipose tissue as a potential protective factor against metabolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-30 years of age at enrollment, who are obese (BMI greater or equal to 30 kg/m2, weight less than 159 kg) and healthy
* Without medications and endocrine/genetic disorders known to affect weight.
* Participants may have insulin resistance, impaired glucose tolerance, dyslipidemia, or hypertension.

Exclusion Criteria:

* Anyone who refuses participation.
* A genetic syndrome or other endocrine disorder known to cause obesity (Prader-Willi, Cushing Syndrome, Leptin deficiency, etc.).
* Use of the following medications: psychotropics, sulphonylurea, thiazolidinediones, insulin, glucocorticoids, anti-neoplastic agents, angiotensin receptor blocker, angiotensin-converting enzyme inhibitors.
* Pregnancy or history of pregnancy.
* Active infectious disease
* History of CVD or stroke during the previous 36 months
* Total cholesterol 300 mg/dl, triglycerides 400 mg/dl
* Blood pressure 140/90 mmHg
* Fasting plasma glucose 126 mg/dl.
* Diabetes mellitus, type 1 or 2.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, obese young adults
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2010-06; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Presence of brown adipose tissue | 2 years

SECONDARY OUTCOMES:
Presence of metabolic dysfunction | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Mihalopoulos, Principal Investigator — University of Utah, Department of Pediatrics, Division of Adolescent Medicine
Locations (1):
- University of Utah, Salt Lake City, Utah, United States